CLINICAL TRIAL: NCT05216692
Title: Effects of a Foot Strengthening Protocol on Foot Strength, Foot Morphological Deformation and Kinetics Parameters : a Monocentric Randomized Controlled Trial
Brief Title: Morphological and Functional Effects of a Foot Strengthening Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: François Fourchet (Other)
Responsible Party: Sponsor-Investigator, François Fourchet, PhD, Physiotherapist. Head of physiotherapy and ergotherapy., La Tour Hospital
Organization: La Tour Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-D0041
Record Dates: First submitted 2021-12-14; First posted 2022-01-31 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Foot Strength Deficit

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The foot strengthening protocol will last 4 weeks with 2 sessions per week and is composed of 3 exercises targeting forefoot and midfoot region strength as well as enhancing plyometric capabilities of the foot complex.
  Interventions: Procedure: La Tour Hospital Foot Strengthening Protocol
- Control group (Active Comparator): The standard literature foot strengthening protocol will last 4 weeks with 3 sessions per week and is composed of one exercise targeting the strength of the foot medial arch.
  Interventions: Procedure: Standard Literature Foot Strengthening Protocol

INTERVENTIONS:
Procedure: La Tour Hospital Foot Strengthening Protocol — First exercise : "NMES forward lean doming". Doming exercise assisted by NMES placed on the IFM. 8 sec of contraction (6 sec rest) moving the trunk forward. 12 repetitions, 3 sets. Progressive increase of the intensity of NEMS during 4 weeks and increase of body load while decreasing the number of repetitions.
  Second exercise : "MTP joint flexion". Isometric MTP joint flexion contractions. 4 contractions of 5 sec (10 sec rest), 3 sets. Progressive increase of the number of MVIC during 4 weeks and of increase body load while keeping the same intensity.
  Third exercise : "Foot-ankle rebound". Multiple jumps with only plantar flexion. Keeping the knee stiff and straight and pushing off the ground with only ankle and MTP plantar flexion by a forefoot contact with the ground. 10 seconds of jump (1 min of rest) during 5 sets. Progressive increase of body load while keeping the same intensity.
  Arms: Experimental group
Procedure: Standard Literature Foot Strengthening Protocol — During the 1st week, the participants will perform the "Short foot exercise" (SFE) during 3 series of 10 repetitions of 5 seconds of contractions in sitting position. 1 minute of rest will be give between series.
  During the 2nd week, the participants will perform the SFE during 3 series of 15 repetitions of 5 seconds of contractions in sitting position. 1 minute of rest will be give between series.
  During the 3rd week, the participants will perform the SFE during 3 series of 15 repetitions of 5 seconds of contractions in standing bipedal position. 1 minute of rest will be give between series.
  During the 4th week, the participants will perform the SFE during 3 series of 15 repetitions of 5 seconds of contractions in standing unipedal position. 1 minute of rest will be give between series.
  The progression of the exercise during the protocol will be based on passing from a sitting position to a unipedal standing position.
  Arms: Control group

SUMMARY:
The principal aim of this study is to investigate the effects of a four-week foot strenghtening protocol combining active voluntary exercises and assisted-active voluntary exercises by neuromuscular electrical stimulation on hallux toe flexion strength in comparison to a standard foot strengthening protocol in a healthy adult recreational active population.

The secondary objectives of the study are to investigate the effects of this protocol on lesser toes flexor strength, foot morphology deformation in one, two and three dimensions and kinetic parameters when walking and running.

ELIGIBILITY:
Inclusion Criteria:

- Level of weekly physical activity (recreational activity and regular non-competitive runners : at least 1 running session per week)

Exclusion Criteria:

* History of pain or episodes of foot or ankle sprains during the past 6 months;
* Foot or leg fractures during the past year;
* Severe deformity of the foot or leg;
* Self-declared disability due to neuromuscular impairment of the lower limbs;
* Neurological or vestibular deficit that could hinder balance (diabetes mellitus, radiculopathie lumbosacral, soft tissue disorder such as Marfan or Ehlers-Danlos syndrome) ;
* Any absolute contraindication to neuromuscular electrical stimulation (NMES) (cardiac pacemaker, epileptic disorders, pregnancy defibrillator);
* Participation in an exercise program specifically designed to strengthen the ankle or foot during the last 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Hallux flexion strength | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Hallux flexion strength will be assessed by a MicroFET2 Handheld Digital Dynamometer in hook lying position. The strength will be normalized by bodyweight (N/kg).

SECONDARY OUTCOMES:
Change in Lesser toe flexion strength | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Lesser toe flexion strength will be assessed by a MicroFET2 Handheld Digital Dynamometer in hook lying position. The strength will be normalized by bodyweight (N/kg).
Change in Foot morphological deformation | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Foot morphological deformation in 1, 2 and 3 dimensions will be assessed thanks to the Arch Height Index Measurement System (AHIMS, JAKTOOL Corporation, Cranberry, NJ) by measuring the change of the total foot length, foot width, truncated foot length, dorsal arch height, navicular height measurements in a sitting position (10% of bodyweight) to a standing position (95% of bodyweight). The percentage of loading during the measurement will be checked by performing the measurement of force platform.
Change in Running and walking kinetics : Time parameters | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Running kinetic parameters when walking and running will be assessed with an instrumented treadmill (Zebris FDM-THQ, ZebrisMedicalGmbH, Germany). The variables collected will be mean contact time (s), mean flight time (s), and the duration (s) on 7-foot regions (heel 1, heel 2, midfoot, forefoot 1, forefoot 2, forefoot 3, toes) will be assessed during 40 seconds of acquisition at self-selected speed during walking and running.
Change in Running and walking kinetics : Force parameters | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Running kinetic parameters when walking and running will be assessed with an instrumented treadmill (Zebris FDM-THQ, ZebrisMedicalGmbH, Germany). The variables collected will be mean vertical force (N) and peak force (N) on 7-foot regions (heel 1, heel 2, midfoot, forefoot 1, forefoot 2, forefoot 3, toes) during 40 seconds of acquisition at self-selected speed during walking and running.
Change in Running and walking kinetics : Distance parameters | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Running kinetic parameters when walking and running will be assessed with an instrumented treadmill (Zebris FDM-THQ, ZebrisMedicalGmbH, Germany). The variables collected will be step length (cm) and step width (cm) during 40 seconds of acquisition at self-selected speed during walking and running.
Change in Running and walking kinetics : Stiffness parameter | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Running kinetic parameters when walking and running will be assessed with an instrumented treadmill (Zebris FDM-THQ, ZebrisMedicalGmbH, Germany). The variable collected will be mean kleg (Kn/m) during 40 seconds of acquisition at self-selected speed during walking and running.
Change in Running and walking kinetics : Frequency parameter | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Running kinetic parameters when walking and running will be assessed with an instrumented treadmill (Zebris FDM-THQ, ZebrisMedicalGmbH, Germany). The variable collected will be step frequency (step/min) during 40 seconds of acquisition at self-selected speed during walking and running.
Change in Running and walking kinetics : Pressure parameter | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Running kinetic parameters when walking and running will be assessed with an instrumented treadmill (Zebris FDM-THQ, ZebrisMedicalGmbH, Germany). The variable collected will be the maximal pressure (N/cm²) on 7-foot regions (heel 1, heel 2, midfoot, forefoot 1, forefoot 2, forefoot 3, toes) during 40 seconds of acquisition at self-selected speed during walking and running.

OTHER OUTCOMES:
Change in Evertor and invertor anke muscles strength | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Evertor and invertor anke muscles strength will be assessed by a MicroFET2 Handheld Digital Dynamometer in supine position and with the ankle in neutral position. The strength will be normalized by bodyweight (N/kg).
Change in Plantarflexor muscles strength | All measures will be collected on both feet 1 week prior the treatment and 1 week after the last intervention session
  Plantarflexor strength will be assessed by using the Heel-Rise Test according to previous recommendations. The maximal repetitions will be keep for the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: François Fourchet, PhD, Principal Investigator — La Tour Hospital, Human Motion Lab
Locations (1):
- Hopital de La Tour, Service de Physiothérapie, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fraser JJ, Hertel J. Effects of a 4-Week Intrinsic Foot Muscle Exercise Program on Motor Function: A Preliminary Randomized Control Trial. J Sport Rehabil. 2019 May 1;28(4):339-349. doi: 10.1123/jsr.2017-0150. Epub 2018 Dec 4. PMID 29364026
- [Result] Kim KM, Croy T, Hertel J, Saliba S. Effects of neuromuscular electrical stimulation after anterior cruciate ligament reconstruction on quadriceps strength, function, and patient-oriented outcomes: a systematic review. J Orthop Sports Phys Ther. 2010 Jul;40(7):383-91. doi: 10.2519/jospt.2010.3184. PMID 20592480
- [Result] Namsawang J, Eungpinichpong W, Vichiansiri R, Rattanathongkom S. Effects of the Short Foot Exercise With Neuromuscular Electrical Stimulation on Navicular Height in Flexible Flatfoot in Thailand: A Randomized Controlled Trial. J Prev Med Public Health. 2019 Jul;52(4):250-257. doi: 10.3961/jpmph.19.072. Epub 2019 Jul 14. PMID 31390688
- [Result] Taddei UT, Matias AB, Ribeiro FIA, Bus SA, Sacco ICN. Effects of a foot strengthening program on foot muscle morphology and running mechanics: A proof-of-concept, single-blind randomized controlled trial. Phys Ther Sport. 2020 Mar;42:107-115. doi: 10.1016/j.ptsp.2020.01.007. Epub 2020 Jan 13. PMID 31962191
- [Result] McKeon PO, Hertel J, Bramble D, Davis I. The foot core system: a new paradigm for understanding intrinsic foot muscle function. Br J Sports Med. 2015 Mar;49(5):290. doi: 10.1136/bjsports-2013-092690. Epub 2014 Mar 21. PMID 24659509
- [Result] Gooding TM, Feger MA, Hart JM, Hertel J. Intrinsic Foot Muscle Activation During Specific Exercises: A T2 Time Magnetic Resonance Imaging Study. J Athl Train. 2016 Aug;51(8):644-650. doi: 10.4085/1062-6050-51.10.07. Epub 2016 Oct 3. PMID 27690528
- [Result] Fourchet F, Kuitunen S, Girard O, Beard AJ, Millet GP. Effects of Combined Foot/Ankle Electromyostimulation and Resistance Training on the In-Shoe Plantar Pressure Patterns during Sprint in Young Athletes. J Sports Sci Med. 2011 Jun 1;10(2):292-300. eCollection 2011. PMID 24149874
- [Result] Gaillet JC, Biraud JC, Bessou M, Bessou P. Modifications of baropodograms after transcutaneous electric stimulation of the abductor hallucis muscle in humans standing erect. Clin Biomech (Bristol). 2004 Dec;19(10):1066-9. doi: 10.1016/j.clinbiomech.2004.03.005. PMID 15531058
- [Result] Fiolkowski P, Brunt D, Bishop M, Woo R, Horodyski M. Intrinsic pedal musculature support of the medial longitudinal arch: an electromyography study. J Foot Ankle Surg. 2003 Nov-Dec;42(6):327-33. doi: 10.1053/j.jfas.2003.10.003. PMID 14688773
- [Result] Soysa A, Hiller C, Refshauge K, Burns J. Importance and challenges of measuring intrinsic foot muscle strength. J Foot Ankle Res. 2012 Nov 26;5(1):29. doi: 10.1186/1757-1146-5-29. PMID 23181771
- [Result] Kelly LA, Kuitunen S, Racinais S, Cresswell AG. Recruitment of the plantar intrinsic foot muscles with increasing postural demand. Clin Biomech (Bristol). 2012 Jan;27(1):46-51. doi: 10.1016/j.clinbiomech.2011.07.013. Epub 2011 Aug 23. PMID 21864955
- [Result] Kelly LA, Lichtwark G, Cresswell AG. Active regulation of longitudinal arch compression and recoil during walking and running. J R Soc Interface. 2015 Jan 6;12(102):20141076. doi: 10.1098/rsif.2014.1076. PMID 25551151
- [Result] Kelly LA, Farris DJ, Lichtwark GA, Cresswell AG. The Influence of Foot-Strike Technique on the Neuromechanical Function of the Foot. Med Sci Sports Exerc. 2018 Jan;50(1):98-108. doi: 10.1249/MSS.0000000000001420. PMID 28902682